CLINICAL TRIAL: NCT05524155
Title: Safety and Efficacy of Sintilimab Combined With Regorafenib and HAIC in Patients With Colorectal Liver Metastasis Who Failed Second-line Therapy
Brief Title: Sintilimab Combined With Regorafenib and HAIC in Patients With Colorectal Liver Metastasis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Principal Investigator, Tongguo Si, associate chief physician, Tianjin Medical University Cancer Institute and Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRHCL
Record Dates: First submitted 2022-08-26; First posted 2022-09-01 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Colorectal Cancer; Liver Metastasis
Keywords: Colorectal Liver Metastasis; Sintilimab; Regorafenib; HAIC
MeSH Terms: conditions — Colorectal Neoplasms | interventions — sintilimab; regorafenib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintilimab Combined With Regorafenib and HAIC (Experimental): Sintilimab Combined With Regorafenib and HAIC
  Interventions: Drug: HAIC; Drug: Sintilimab; Drug: Regorafenib

INTERVENTIONS:
Drug: HAIC — hepatic arterial infusion (HAI) of oxaliplatin, fluorouracil/leucovorin (FOLFOX) treatment
  Other Names: Hepatic Artery Infusion Chemotherapy
Drug: Sintilimab — 200mg IV d1,Q3W
  Other Names: IBI308
Drug: Regorafenib — 80mg/day,PO,QD,d1～21,Q4W

SUMMARY:
To evaluate the safety and efficacy of sintilimab combined with regorafenib and HAIC in patients with colorectal liver metastasis who failed second-line therapy

ELIGIBILITY:
Inclusion Criteria:

* Sign written informed consent before performing any trial related procedures
* ≥ 18 years old
* Histologically or cytologically proven unresectable metastatic colorectal cancer with liver metastases (AJCC 8th IV)
* Intolerance to second-line therapy, or disease progression during or after second-line therapy (RECIST V1.1)
* At least one radiographically measurable lesion, according to the RECIST V1.1 criteria
* Patients with asymptomatic brain metastases or stable symptoms after local treatment were allowed to enroll if they met the following criteria:

  * Measurable lesions outside the central nervous system
  * No central nervous system symptoms, or symptoms not worsened for at least 2 weeks
  * No glucocorticoid therapy was required or glucocorticoid therapy was discontinued within 7 days before the first study drug administration
* Palliative radiation therapy (including craniocerebral radiation for symptomatic brain metastases) was permitted, provided that the radiation had ended at least 1 week before enrollment and that the radiotherapy-related toxicity had recovered to grade 1 or less (CTCAE 5.0, except alopecia).
* ECOG PS scores 0-1
* The expected survival time was >3 months
* Sufficient organ functions, the subjects need to meet the following laboratory indicators:

  * ANC ≥1.5×10^9/L without the use of granulocyte colony-stimulating factor in the last 14 days
  * Platelets ≥90×10^9/ without blood transfusion in the past 14 days
  * Hemoglobin >9g/dL without blood transfusion or erythropoietin use in the past 14 days
  * Total bilirubin ≤1.5× upper limit of normal (ULN); Or total bilirubin >ULN but direct bilirubin ≤ ULN
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) in ≤2.5×ULN (ALT or AST ≤5×ULN allowed in patients with liver metastases)
  * Serum creatinine ≤ 1.5 × ULN and creatinine clearance rate (calculated by Cockcroft-Gault formula) ≥ 60 ml/min
  * Good coagulation function, defined as international normalized ratio (INR) or prothrombin time (PT) ≤1.5 × ULN
  * Normal thyroid function, defined as thyroid stimulating hormone (TSH) within normal limits. If the baseline TSH was outside the normal range, subjects with total T3 (or FT3) and FT4 within the normal range could also be enrolled
  * The myocardial zymogram is within the normal range (if the investigator comprehensively determines that the simple laboratory abnormality is not of clinical significance, it is also allowed to be enrolled)
* Pregnancy test negative and use birth control

Exclusion Criteria:

* Previous treatment with regorafenib
* Previous treatment with anti-PD-L1, anti-PD-L2 drugs, or other drugs that stimulates or synergistically inhibits T-cell receptors (e.g., CTLA-4, OX-40, CD137)
* Symptomatic or high risk of obstruction, bleeding, perforation, pneumonia (including noncommunicable pneumonia with previous hormonal therapy and pneumonia in patients receiving treatment)
* Malignancy other than colorectal cancer diagnosed within 5 years before the first dose (excluding radical basal cell carcinoma of the skin, squamous carcinoma of the skin, and/or carcinoma in situ after radical resection)
* currently participating in an interventional clinical study treatment, or has received another study drug or used a study device within 4 weeks prior to the first dose
* Systemic systemic therapy with proprietary Chinese medicine or immunomodulatory agents (including thymosin, interferon, and interleukin, except for local use to control pleural effusion) with anti-tumor indications was received within 2 weeks before the first dose
* Active autoimmune disease requiring systemic therapy occurred within 2 years before the first dose. Alternative therapies (e.g., thyroxine, insulin, or physiologic glucocorticoids for adrenal or pituitary insufficiency) are not considered systemic therapy
* Receiving systemic glucocorticoid therapy (excluding intranasal, inhaled, or other local glucocorticoids) or any other form of immunosuppressive therapy within 7 days before the first dose; Physiological doses of glucocorticoids (≤10 mg/day or equivalent prednisone) are permitted
* Blood transfusion within 7 days before the first dose
* Clinically uncontrollable pleural effusion/abdominal effusion
* Known allogeneic organ transplantation (excluding corneal transplantation) or allogeneic hematopoietic stem cell transplantation
* Known allergy to the active ingredient or excipient of the study drug
* Not fully recovered from toxicity and/or complications caused by any intervention (≤ grade 1 or baseline, excluding fatigue or alopecia) before starting treatment
* HIV 1/2 antibody positive
* Untreated active hepatitis B, subjects who met the following criteria could also be enrolled:

  * HBV viral load <1000 copies/ml (200 IU/ml) before the first dose, subjects should receive anti-HBV therapy to avoid virus reactivation throughout the study
  * Subjects with anti-HBC (+), HBsAg (-), anti-HBs (-), and HBV viral load (-) did not require prophylactic anti-HBV therapy, but did require close monitoring for viral reactivation
* Active HCV-infected
* Received live vaccine within 30 days prior to the first dose，Inactivated virus vaccines for injectable use against seasonal influenza are permitted up to 30 days before the first dose，live attenuated influenza vaccines administered intranasally not allowed
* Pregnant or lactating woman
* With any severe or uncontrolled systemic disease
* Other conditions that the subjects are not suitable to participate in this study according to the judgment of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AEs) | up to 24 months
  Defined as the proportion of patients with AE, treatment-related AE (TRAE), immune-related AE (irAE), serious adverse event (SAE), assessed by NCI CTCAE v5.0
Overall response rate ( ORR) | up to 24 months
  Defined as proportion of patients who have a best response of CR or PR

SECONDARY OUTCOMES:
Disease control rate (DCR) | up to 24 months
  Defined as proportion of patients who have a best response of CR, PR or SD
Duration of response (DoR) | up to 24 months
  Defined as the time from first confirmed response (CR or PR) to the date of the first documented tumor progression or death due to any cause, whichever occurs first.
Progression free survival (PFS) | up to 28 months
  Defined as the time from enrollment to disease progression or death, whichever occurs first
Overall survival (OS) | up to 28 months
  Defined as the time from the date of treatment start to the date of death